CLINICAL TRIAL: NCT01299428
Title: Evaluation of the Cerebral Oxygenation With Near Infrared Spectrophotometry (NIRS) at the Hypernatremic Dehydration in Newborn
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Zekai Tahir Burak Maternity Teaching Hospital, Zekai Tahir Burak Maternity Teaching Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 5
Record Dates: First submitted 2011-02-17; First posted 2011-02-18 (Estimated); Last update posted 2011-02-18 (Estimated); Status verified 2011-02

CONDITIONS: HYPERNATREMIA
Keywords: CEREBRAL OXYGENATION; HYPERNATREMİA; NEWBORN; NA VALUES
MeSH Terms: conditions — Hypernatremia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cerebral oxygenation (Active Comparator)
  Interventions: Device: INVOS 5100

INTERVENTIONS:
Device: INVOS 5100 — INVOS 5100 IS AN EQUIPMENT THAT MEASURED CEREBRAL OXYGENATION WITH NEAR INFRARED SPECTROPHOTOMETRY METHOD.

SUMMARY:
The aim of the study is to evaluate cerebral oxygenation with Near infrared spectrophotometry (NIRS) at the hypernatremic dehydration in newborns.

ELIGIBILITY:
Inclusion Criteria:

* gestation week > 37 ve Na >150 mg/dl
* Dehydration

Exclusion Criteria:

* Sepsis
* Intracranial Haemorrhagia
* Congenital Cardiac Diseases

Ages: 1 Day to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-05 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
CEREBRAL OXYGENATION | 3 MONTHS
  NIRS METHODS

SECONDARY OUTCOMES:
NEURODEVELOPMENT | 12-18 MONTHS
  NEURODEVELOPMENT EVALUATION

CONTACTS AND LOCATIONS:
Locations (1):
- Zekai Tahir Burak Maternity Teaching Hospital, Ankara, Samanpazarı, Turkey (Türkiye)